CLINICAL TRIAL: NCT03288454
Title: Phase 2 Placebo-Controlled, Single-Site, Single-Blind Study of Apixaban Reversal by Ciraparantag as Measured by WBCT
Brief Title: Phase 2 Study of Apixaban Reversal by Ciraparantag as Measured by WBCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PER977-02-011
Record Dates: First submitted 2017-09-14; First posted 2017-09-20 (Actual); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Ciraparantag; PER977; Apixaban; Whole Blood Clotting Time (WBCT)
MeSH Terms: interventions — PER977; apixaban

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): ciraparantag (60 mg)
  Interventions: Drug: Ciraparantag; Drug: Apixaban
- Cohort 2 (Experimental): ciraparantag (120 mg)
  Interventions: Drug: Ciraparantag; Drug: Apixaban
- Cohort 3 (Experimental): ciraparantag (30 mg)
  Interventions: Drug: Ciraparantag; Drug: Apixaban
- Placebo (Placebo Comparator): placebo (saline for injection)
  Interventions: Drug: Placebo; Drug: Apixaban

INTERVENTIONS:
Drug: Ciraparantag — Ciraparantag (administered over 10 minutes)
  Other Names: PER977; AMAG 977
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Placebo — Saline for injection
  Other Names: PBO
  Arms: Placebo
Drug: Apixaban — Apixaban 10mg given twice daily (q12h)

SUMMARY:
This study is a randomized, single-blind, placebo-controlled study to assess the efficacy and safety of ciraparantag administered to healthy volunteers anticoagulated with apixaban measuring clotting times using Whole Blood Clotting Time (WBCT).

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled assessment of the efficacy and safety of ciraparantag administered to healthy volunteers measuring clotting times using WBCT as determined by the manual testing method. All subjects will undergo screening up to 36 days prior to enrollment.

All enrolled subjects are to receive 10 mg apixaban orally for 3.5 days (every 12 hours on Days 1-3 and once on the morning of Day 4). On Day 4, subjects who achieve sufficient anticoagulation (WBCT ≥20% above baseline) are randomized and will receive a single dose of study drug (ciraparantag or placebo) intravenously (IV) approximately 3 hours after the apixaban dose, followed by serial testing of manual WBCT.

Subjects are enrolled sequentially into 3 ciraparantag dose cohorts. There will be a safety review after completion of treatment in one cohort and prior to initiation of treatment in the subsequent cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 50 to 75 years, inclusive
2. Laboratory tests (chemistry, hematology and coagulation assessments) and urinalysis performed during screening up to 36 days prior to administration of study treatment deemed not clinically significant by the principal investigator.
3. No clinically significant findings on 12-lead electrocardiogram (ECG) performed during screening
4. Body mass index (BMI) 18 to ≤ 32 kg/m2, inclusive
5. Male subjects agree to use appropriate contraception (i.e., latex condom with spermicide) in addition to their partner using an acceptable form of contraception (e.g., diaphragm, cervical cap, intrauterine device, hormonal contraceptives, surgical sterilization or post-menopausal), when engaging in sexual activity during the course of the study. Moreover, male subjects should not donate sperm or attempt to impregnate a partner during the course of the study and for a period of 12 weeks following discharge from the study.
6. Female subjects must have negative pregnancy tests at screening and check-in AND: be surgically sterile at least 6 months prior to the first dose (with documentation of hysterectomy, bilateral oophorectomy, bilateral salpingectomy, bilateral tubal ligation/tubal occlusion); OR post-menopausal (no menstruation for a minimum of 12 months and confirmed by follicle stimulating hormone [FSH] of ≥ 40 mIU/ml and serum estradiol < 30 pg/ml at screening and check-in); OR if of childbearing potential, must be using an acceptable method of contraception such as an intrauterine device (IUD), implant or contraceptive injection, or two forms of the following (e.g., diaphragm, cervical cap, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge) for the last three months. All females must agree to continue to use their method of birth control for the duration of the study and for a minimum of one complete menstrual cycle from the study
7. Subjects who have participated in a prior study of ciraparantag must have been discharged from the study a minimum of 1 month prior to the planned treatment.
8. Subjects must understand and agree to comply with the requirements of the study and they must be willing to sign the informed consent form indicating voluntary consent to participate in the study prior to initiation of screening or study-related activities -

Exclusion Criteria:

1. History or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine, neurologic, infectious, gastrointestinal (including gallbladder disease or surgery), hematologic, or oncologic disease as determined by screening history, physical examination, laboratory test results or 12-lead ECG assessment. History or current evidence of liver function tests greater than 50% of the upper limit of normal (ULN) or renal function tests (serum creatinine) greater than 1.5 mg/dl and based on PI discretion. History or current evidence of QTc (QTcF) greater than normal (450 msec for males or 470 msec for females).
2. History of unexplained syncope
3. History of major bleeding, trauma, or surgical procedure of any type based on PI discretion
4. Vaginal delivery within six months prior to screening
5. History of peptic ulcer, gastrointestinal bleeding (including hematemesis, melena, rectal bleeding) within one year prior to screening
6. Long standing history of bleeding episodes such as epistaxis, bruising or gingival bleeding or if not long standing, within 1 month prior to screening
7. Personal or family history of clotting disorder or abnormality, excessive bleeding, joint hematoma, thrombovascular disease or any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, or history of thrombocytopenia
8. Females with a history of dysfunctional uterine bleeding who have not undergone hysterectomy, including history of menorrhagia (heavy menstrual bleeding), menometrorrhagia or polymenorrhea
9. Smokers or use of tobacco and/or nicotine containing products within 3 months prior to dosing as determined by the subject's verbal history
10. Pregnant or breast-feeding
11. Males with a history of hormone therapy within 3 months prior to screening
12. Taking any type of chronic medication (including vitamin, nutritional and herbal supplements) for more than 14 consecutive days within the 4 weeks prior to study entry (use of hormonal contraceptives is acceptable except for oral contraceptives)
13. Positive serologic test for human immunodeficiency virus (HIV), Hepatitis C virus antibody (HCV-Ab), or Hepatitis B surface antigen (HBsAg)
14. Donation of blood or blood products within 56 days prior to screening
15. Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
16. Active drug or alcohol dependence within the prior 12 months or any condition that, in the opinion of the Investigator, would interfere with adherence to study protocol
17. Allergic to apixaban

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Frontage Clinical Services Inc., Secaucus, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One study site in the US enrolled subjects between August 2017 and August 2019.
Pre-assignment Details: 60 subjects enrolled; 49 subjects were randomized and eleven subjects were not randomized. Of the 11 subjects not randomized, 9 did not achieve a sufficient level of anticoagulation per protocol and 2 had adverse events (AEs) during apixaban administration causing discontinuation (headache and electrocardiogram abnormal).
Groups:
- Placebo: Subjects received 10 mg apixaban twice daily on Days 1-3 and once on the morning of Day 4. On Day 4, approximately 3 hours after last apixaban dose, a single IV dose of saline for injection (placebo) was administered.
- Ciraparantag 30mg: Subjects received 10 mg apixaban twice daily on Days 1-3 and once on the morning of Day 4. On Day 4, approximately 3 hours after last apixaban dose, a single IV dose of 30 mg ciraparantag was administered.
- Ciraparantag 60 mg: Subjects received 10 mg apixaban twice daily on Days 1-3 and once on the morning of Day 4. On Day 4, approximately 3 hours after last apixaban dose, a single IV dose of 60mg ciraparantag was administered.
- Ciraparantag 120 mg: Subjects received 10 mg apixaban twice daily on Days 1-3 and once on the morning of Day 4. On Day 4, approximately 3 hours after last apixaban dose, a single IV dose of 120mg ciraparantag was administered.
Period: Overall Study
Arm/Group | Placebo | Ciraparantag 30mg | Ciraparantag 60 mg | Ciraparantag 120 mg
Started | 13 | 12 | 12 | 12
Completed | 13 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population, defined as all subjects who receive at least 1 administration of investigational product (ciraparantag or placebo), was used for all baseline measures except for WBCT, which uses the Pharmacodynamic Population. These populations differ only in the placebo group which has 12 subjects for WBCT baseline measure.
Groups:
- Ciraparantag 30 mg: Subjects received 10 mg apixaban twice daily on Days 1-3 and once on the morning of Day 4. On Day 4, approximately 3 hours after last apixaban dose, a single IV dose of 30mg ciraparantag was administered.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg | Total
Number analyzed (Participants) | 13 | 12 | 12 | 12 | 49
Age, Customized [Mean (Standard Deviation); unit: years] | 57.2 (6.90) | 55.8 (5.72) | 54.4 (3.87) | 53.9 (4.13) | 55.4 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 1 | 11
  Male | 10 | 8 | 9 | 11 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 4 | 3 | 14
  Not Hispanic or Latino | 8 | 10 | 8 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 3 | 9 | 21
  White | 8 | 7 | 8 | 3 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.36 (3.70) | 26.22 (3.03) | 26.40 (2.47) | 26.59 (2.98) | 26.66 (3.03)
Baseline Whole Blood Clotting Time (WBCT, manual method) [Mean (Standard Deviation); unit: minutes] — Population: Pharmacodynamic Population included all subjects who received administration of ciraparantag/placebo and provided at least one on-treatment WBCT measurement without protocol deviations with potential to affect these measurements.
  minutes
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
    (all) | 7.4 (0.29) | 7.7 (0.33) | 7.3 (0.26) | 7.5 (0.33) | 7.5 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: Subjects Achieving Complete Reversal of Anticoagulation (WBCT is ≤ 110% of Baseline)
Description: Complete reversal is achieved if WBCT (manual method) is ≤ 110% of baseline at any post-baseline time point up to and including 1 hour following ciraparantag/PBO administration
Time Frame: Within 1 Hour
Population: Pharmacodynamic population: all subjects who receive administration of study drug and provide at least one on-treatment whole blood clotting time measurement without protocol deviations with potential to affect these measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 2 | 9 | 12 | 12

2. Primary Outcome: Subjects Achieving Complete and Sustained Reversal of Anticoagulation (WBCT is ≤115% of Baseline)
Description: Complete and sustained reversal of anticoagulation is achieved for a subject if WBCT (manual method) is ≤ 115% of baseline at all time points between 1 and 5 hours (inclusive) following ciraparantag/placebo administration.
Time Frame: Between 1 and 5 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 4 | 10 | 12 | 12

ADVERSE EVENTS:
Time Frame: All AEs occurring after the subject signed the informed consent through the last study visit (follow-up phone call occurring 7 to 10 days following ciraparantag/PBO administration), whether observed by the Investigator or reported by the subject, were collected. SAEs occurring up to 30 calendar days post treatment were collected.
Groups:
- Enrolled But Not Randomized Participants: Subjects received 10 mg apixaban twice daily on Days 1-3 and once on the morning of Day 4. On Day 4, the subjects were not randomized due to WBCT below required threshold or subject discontinued early due to adverse event.
Arm/Group | Placebo | Ciraparantag 30 mg | Ciraparantag 60 mg | Ciraparantag 120 mg | Enrolled But Not Randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/12 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 1/13 | 4/12 | 6/12 | 8/12 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Ciraparantag 30 mg (N=12) | Ciraparantag 60 mg (N=12) | Ciraparantag 120 mg (N=12) | Enrolled But Not Randomized Participants (N=11)
Hot flush (Vascular disorders) | 0 | 1 | 5 | 2 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 3 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Hypoesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT03288454/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT03288454/SAP_001.pdf